CLINICAL TRIAL: NCT03752827
Title: A Prospective, Double-Blinded, Multi-Center Pivotal Trial of Autologous Adult Adipose-Derived Regenerative Cell Injection Into Chronic Partial-Thickness Rotator Cuff Tears
Brief Title: Autologous Adult Adipose-Derived Regenerative Cell Injection Into Chronic Partial-Thickness Rotator Cuff Tears
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC-002
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Tendinitis
Keywords: rotator cuff tear; adipose-derived regenerative cells; adipose-derived stem cells; partial rotator cuff tears; corticosteroid
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: It is a double-blinded trial in which the subject, post-procedural investigator and imaging core laboratory radiologists are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adipose Derived Regenerative Cells (Experimental): Adipose-derived regenerative cell injection into the area of the supraspinatus tendon tear
  Interventions: Device: Adipose Derived Regenerative Cells
- Corticosteroid (Active Comparator): Subjects in the active control arm will receive a corticosteroid injection into the subacromial space using ultrasound (US) guidance.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Device: Adipose Derived Regenerative Cells — Adipose-derived regenerative cells isolated with the Transpose Ultra system
  Arms: Adipose Derived Regenerative Cells
Drug: Corticosteroid — Corticosteroid injection into subacrominal space
  Arms: Corticosteroid

SUMMARY:
The purpose of this investigation is to evaluate the safety and superior effectiveness in functional improvement in patients with partial-thickness rotator cuff tears (PTRCTs) after the administration of a single injection of adipose-derived regenerative cells (ADRCs) into the partial-thickness rotator cuff tear compared to the administration of a single corticosteroid injection into the associated subacromial space.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, randomized, active-controlled, multi-site, pivotal safety and superior effectiveness study in patients with symptomatic partial-thickness rotator cuff tears comparing a single ADRC injection generated with the Transpose® RT system into the supraspinatus tendon and surrounding area to standard-of-care (SOC) corticosteroid injection into the subacromial bursa.

Up to 20 U.S. centers will be initiated to enroll in the study. 246 subjects assigned to two randomization arms will be enrolled: an adipose-derived regenerative cell (ADRC) injection arm (ADRC treatment arm) and the SOC corticosteroid injection arm (active control arm). All subjects will be randomly assigned to ADRC treatment or active control arms in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 30-75 years of age (inclusive).
2. Subjects have a minimum of three (3) months of clinical symptoms consistent with a partial-thickness rotator cuff tear including but not limited to pain, muscle weakness, or limited active range of motion (AROM).
3. Subjects have > 70% passive range of motion (PROM) of the index shoulder.
4. Subjects have a baseline VAS - Pain score of ≥ 30 mm.
5. Subjects have a partial-thickness rotator cuff tear, defined as ≥25% partial-thickness tear of the supraspinatus tendon on a 1.5 Tesla (1.5T) or a 3 Tesla (3T) MRI within the last 3 months, as determined by the Investigator.
6. Subjects can give appropriate consent.

Exclusion Criteria:

1. Age < 30 or > 75.
2. Subject has an insufficient amount of subcutaneous tissue to allow recovery of 100 milliliters (mL) of adipose tissue.
3. Subjects who have received a corticosteroid injection in the index subacromial bursa within the last 3 months.
4. Subjects who have received more than one (1) previous corticosteroid injections or any biologic treatment in the index subacromial bursa within the past 6 months.
5. Subjects with severe arthrosis of the glenohumeral or acromioclavicular joint.
6. Subjects with a full-thickness tear of the rotator cuff.
7. Subjects who have undergone major surgery on the affected shoulder meeting one of the following criteria:

   * Performed as treatment for (or required manipulation of) the rotator cuff. Examples include, but are not limited to, subacromial decompression, rotator cuff repair, SLAP repair, arthroplasty and fracture fixation with implants that involve or penetrate the rotator cuff; OR
   * Performed using implants that interfere with MR visualization and/or evaluation of the supraspinatus tendon (e.g., biceps tenodesis); OR
   * Performed in/on the glenohumeral joint, subacromial space, or acromioclavicular joint within the last 3 years (e.g. soft tissue Bankart repairs performed >3 years ago may still qualify).

   NOTE: This exclusion criterion does not apply to minor soft tissue procedures with short recovery periods that do not involve musculoskeletal structures (e.g., lipoma excision).
8. Subjects who were diagnosed with or treated for adhesive capsulitis of the index shoulder within the last 5 years.
9. Subjects with current cervical radiculopathy impacting the index shoulder.
10. Subjects who require the use of index arm for ambulation or mobilization via wheelchair, walker, crutches or cane.
11. Subjects with any contraindication to MRI scan according to MRI guidelines, or who are unwilling to undergo MRI procedures.
12. Subjects whose pain behavior or pain medication usage is, in the opinion of the Investigator, out of proportion to the underlying clinical condition or could interfere with the study- required assessments.
13. Subjects with a history of systemic malignant neoplasms within the last 5 years.
14. Subjects with biopsy-proven, malignant or local neoplasm within the last 6 months or any history of local neoplasm at the site of administration (on the affected arm), excluding basal cell carcinoma.
15. Subject is receiving immunosuppressant therapy or has a known immunologic or severe autoimmune disease that requires chronic systemic immunosuppressive or immunomodulatory therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, rheumatoid arthritis, etc.). [Note: Topical or inhaled corticosteroids are permitted.]
16. Subject is on an active regimen of chemotherapy or radiation- based treatment.
17. Subjects with an allergy to sodium citrate or any "caine" type of local anesthetic.
18. Subject is pregnant or breastfeeding or plans to become pregnant in the next 12 months.
19. Subjects with clinically significant abnormal Lab tests (i.e. basic metabolic panel (BMP) or equivalent (e.g. CHEM-7), complete blood count (CBC), Liver function tests (LFTs), and prothrombin time/international normalized ratio (PT/INR)) as interpreted by the Investigator.

21. Subjects with a history of a bleeding diathesis or coagulopathy

22. Subject is, in the opinion of the Investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. Examples include the inability of the subject to complete patient-reported outcome instruments (PROs) and the inability of the Investigator to perform the injection procedure properly because of anatomic limitations of the subject.

23. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint. (Noninterventional observational studies are not exclusionary.)

24. Subject 1) is a litigant in a civil suit that could affect the subject's ability to complete the study related activities or 2) is a defendant in a criminal case or 3) has an active workman's compensation case in progress.

25. Subject is part of a vulnerable population who, in the judgment of the Investigator, is unable to give informed consent for reasons of incapacity, immaturity, adverse personal. circumstances or lack of autonomy. This may include: individuals with a mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

26. Uncooperative subjects or those with neurological/psychiatric disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Pain: VAS | 24 weeks
  ≥ 14-millimeter (mm) improvement in Visual Analog Scale (VAS)
Improvement or no worsening in supraspinatus strength | 24 weeks
  supraspinatus strength on the MRC Muscle Scale compared to baseline For supraspinatus strength on the MRC Muscle Scale compared to baseline
  • For subjects with normal supraspinatus strength (MRC Muscle Scale = 5] at baseline: no worsening in supraspinatus strength on the MRC Muscle Scale compared to baseline

SECONDARY OUTCOMES:
Percentage of subjects who demonstrate ≥ 14 mm improvement in VAS | 24 weeks
  Pain score compared to baseline at 24 weeks
Percentage of subjects who demonstrate improvement or no worsening of supraspinatus strength on the MRC Muscle Scale | 24 weeks
  Supraspinatus strength on the MRC Muscle Scale compared to baseline at 24 weeks
Mean improvement in VAS - Pain score | 12 and 24 weeks
  VAS pain score compared to baseline
Mean improvement in WORC score | 12 and 24 weeks
  WORC score compared to baseline
Percentage of subjects who demonstrate a ≥ 1-grade improvement in supraspinatus strength on the MRC Muscle Scale | 24 weeks
  Supraspinatus strength on the MRC Muscle Scale compared to baseline at 24 weeks.

OTHER OUTCOMES:
Mean improvement in Rand Short Form-36 score | 24 weeks
  Rand Form-36 score compared at baseline
Measurement of subject satisfaction with treatment on a VAS scale (VAS - Satisfaction) | 24 weeks
  VAS satisfaction score improvement
Measurement of EuroQoL-5D-5L (EQ-5D-5L) | 24 weeks
  EuroQoL -5D-5L score
Measurement of Shoulder Activity Level | 24 weeks
  Recording shoulder activity level
Measurement of shoulder motion (forward elevation, shoulder abduction in the plane of the scapula) | 24 weeks
  As determined by goniometer

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Arizona Research Center, Phoenix, Arizona
  - Biosolutions Clinical Research Center, La Mesa, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Sports and Orthopedic Center, Coral Springs, Florida
  - Universal Axon Clinical Research, Doral, Florida
  - Shrock Clinical Research, Fort Lauderdale, Florida
  - Andrews Institute for Orthopaedics and Sports Medicine, Gulf Breeze, Florida
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Sanford Medical Center, Fargo, North Dakota
  - Sanford Orthopedic Clinic/Research, Sioux Falls, South Dakota
  - HD Research, Houston, Texas
  - Texas Plastic Surgery, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No